CLINICAL TRIAL: NCT00708955
Title: Evaluation and Treatment Protocol for Potential Research Participants With Ocular Diseases
Brief Title: Evaluation and Treatment of People With Eye Diseases
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080169; 08-EI-0169
Record Dates: First submitted 2008-07-02; First posted 2008-07-03 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2017-07-12

CONDITIONS: Eye Diseases
Keywords: Evaluation and Treatment; Eye Diseases
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This study will evaluate and provide standard treatments for people with various eye conditions. It will provide a resource for enrollment into new research protocols throughout the Eye Institute and will allow institute specialists the opportunity to maintain their expertise and gain additional knowledge of the course of various eye disorders. The information obtained will allow for the evaluation of standard treatments and may lead to ideas for future research.

People with diagnosed or undiagnosed eye disease and first-degree relatives of people with a genetic or developmental eye disease may be eligible for this study. Participants are evaluated and treated in the National Eye Institute. Blood or other tissue samples (e.g., urine, stool, hair, saliva or cheek swab) may be collected for future laboratory studies.

DETAILED DESCRIPTION:
The National Eye Institute (NEI) is conducting a study to evaluate and provide standard treatment to participants with various diagnosed and undiagnosed ocular conditions.

Objectives: The primary objective of this protocol is to provide a reservoir of patients for enrollment into new research protocols throughout the NEI laboratories. Evaluating and treating participants will allow the NEI specialists to maintain their expertise and gain additional knowledge of the course of various eye disorders. The information obtained will allow for the evaluation of standard treatments of the studied eye diseases. This understanding may lead to ideas for future protocols. In some cases, blood or other biologic samples (including tear fluid, urine, saliva, hair, stool or a cheek swab) will be obtained for future laboratory studies.

Study Population: The number of participants to be enrolled has no logical upper limit, but will be set to 5,000 patients with ocular diseases and their unaffected first-degree relatives.

Design: This is an observational natural history study of multiple ocular diseases and their progression and physiology.

Outcome Measures: No formal outcomes will be measured; however the clinical assessments of enrolled participants can be used to measure the response to standard treatment. In addition, DNA samples obtained may be used to identify and verify causative mutations, which may help establish pathogenic mechanisms and genotype-phenotype correlations.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants will be eligible if they:

* Have either a diagnosed or undiagnosed eye disease, OR are an unaffected first-degree relative of a participant with a genetic or developmental eye disease.
* Have the ability to understand and sign an informed consent or have a parent/legal guardian to do so if they are minor children.

EXCLUSION CRITERIA:

Participants will not be eligible if they:

* Are unable or unwilling to give informed consent.
* Are unwilling or unable to be followed as clinically indicated.
* Have a systemic disease that compromises the ability to provide adequate ophthalmologic examination or treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2164 (Actual)
Dates: Start 2008-06-25; Study Completion 2017-07-12

CONTACTS AND LOCATIONS:
Overall Officials: Rachel J Bishop, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States